CLINICAL TRIAL: NCT07031141
Title: Diabetes Foot Africa Region Registry
Acronym: (D-FAR)
Status: Not yet recruiting | Type: Observational
Sponsor: Getz Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: GETZ-DF-01-24
Record Dates: First submitted 2025-03-27; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
D-FAR is to gather robust data on the clinical characteristics, management, and outcomes of patients with diabetic foot complications to enhance understanding, reduce complications, and improve patient care. This will include insights into the prevalence of risk factors, adherence to treatment protocols, and the effectiveness of interventions aimed at reducing the incidence of amputations and other adverse outcomes.

DETAILED DESCRIPTION:
Among the various complications, those related to diabetic foot disease are associated with the highest morbidity and mortality. Diabetic foot problems are characterized by infection, ulceration and/or destruction of deep tissue in the foot and are usually associated with neurological abnormalities and varying degrees of peripheral arterial disease (PAD) in the lower limb. the purpose of collect comprehensive data on the clinical features, management strategies, and outcomes of patients with diabetic foot complications.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients
2. Residents of participating African countries.
3. Diagnosed with diabetic foot complications (e.g., ulcers, gangrene, infection, ischemia).
4. Patients with a history of foot ulcers or amputations due to diabetes.
5. High-risk patients with peripheral neuropathy and/or peripheral arterial disease.

Exclusion Criteria:

1. Non-diabetic foot complications.
2. Acute traumatic injuries unrelated to diabetes.
3. Patients unwilling to provide informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: African population
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of Subjects Achieving Complete Wound Healing | Assessed at 3, 6, and 12 months post-enrollment
  Percentage of patients with diabetic foot ulcers who achieve complete wound closure without discharge or infection as recorded during follow-up visits.
  Defined as complete epithelialization of the diabetic foot ulcer with no discharge or infection as assessed during clinical follow-up.
Proportion of Subjects Undergoing Amputation Due to Diabetic Foot Ulcer | Up to 12 months from enrollment
  Number of subjects requiring surgical amputation (minor or major) of the affected foot during the follow-up period

SECONDARY OUTCOMES:
Time Taken for Diabetic Foot Ulcer to Heal | Up to 12 months from enrollment
  Duration (in days) from initial presentation to confirmed complete healing of the ulcer.
Change in SINBAD Score Over Time | Baseline, 3, 6, and 12 months
  SINBAD scores will be measured at baseline and during follow-up to assess changes in wound severity.
  SINBAD is an acronym based on six parameters (Site, Ischemia, Neuropathy, Bacterial infection, Area, and Depth) Scale Range: 0 to 6 Directionality: Higher scores indicate worse outcomes (i.e., more severe diabetic foot ulcer characteristics and higher risk of complications such as non-healing, infection, amputation, or death).
  Interpretation:
  0-1: Mild ulcer, lower risk
  2-3: Moderate ulcer, intermediate risk
  4-6: Severe ulcer, high risk
All-Cause Mortality Among Subjects with Diabetic Foot Ulcers | Up to 12 months from enrollment
  Number and percentage of subjects who expire during the study period, regardless of cause.
Proportion of Subjects with Peripheral Neuropathy and Peripheral Arterial Disease | At baseline
  Presence of peripheral neuropathy and peripheral arterial disease (PAD) in subjects with diabetic foot ulcers based on clinical exam.Can be determined by clinical signs such as loss of protective sensation, absence of pedal pulses, decrease vascularity

CONTACTS AND LOCATIONS:
Overall Officials: Zulfiqarali G Abbas, MBBS, MMed, DTM&H, Principal Investigator — D-Foot International

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abbas ZG, Boulton AJM. Diabetic foot ulcer disease in African continent: 'From clinical care to implementation' - Review of diabetic foot in last 60 years - 1960 to 2020. Diabetes Res Clin Pract. 2022 Jan;183:109155. doi: 10.1016/j.diabres.2021.109155. Epub 2021 Nov 24. PMID 34838640
- [Background] Naemi R, Chockalingam N, Lutale JK, Abbas ZG. Predicting the risk of future diabetic foot ulcer occurrence: a prospective cohort study of patients with diabetes in Tanzania. BMJ Open Diabetes Res Care. 2020 May;8(1):e001122. doi: 10.1136/bmjdrc-2019-001122. PMID 32371531
- [Background] Bak JCG, Serne EH, Kramer MHH, Nieuwdorp M, Verheugt CL. National diabetes registries: do they make a difference? Acta Diabetol. 2021 Mar;58(3):267-278. doi: 10.1007/s00592-020-01576-8. Epub 2020 Aug 8. PMID 32770407
- See also: ocuses on strategies to prevent foot ulcers, including patient education, regular foot examinations, and appropriate footwear.Provides recommendations on relieving pressure (offloading) from foot ulcers to promote healing. — http://iwgdfguidelines.org/guidelines-2019/